CLINICAL TRIAL: NCT03516864
Title: Assessment of Tissue Oxygenation Using Multispectral Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 18-
Record Dates: First submitted 2018-03-08; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus
Keywords: tissue oxygenation; near-infrared; diabetic foot ulcer (DFU); diabetes; vascularity
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MIMOSA Imager — The MultIspectral MObile tiSsue Assessment (MIMOSA) Imager acquires digital images to calculate anatomical details of chronic wounds (e.g. diameter, surface area, and perimeter). The device can be worn from a lanyard, and clips onto a smartphone, using natural ambient lighting to capture images of a wound. The MIMOSA also uses up to 6 near-infrared LEDs to illuminate tissue with different wavelengths of light to assess tissue oxygenation.
Device: Kent Camera — The Food and Drug Administration (FDA) has previously approved a near-infrared device called the Kent camera for the assessment of tissue oxygenation.

SUMMARY:
In Canada, the age-standardized prevalence of diabetes is on the rise (increasing from 3.3% in 1998/99 to 5.6% in 2008/2009 Public Health Agency of Canada (July 2011)) and is almost 1 in 10 globally. One of the most devastating complications of diabetes is the loss of a limb, (also known as lower extremity amputation, or LEA) due to complications resulting from a diabetic foot ulcer (DFU). Diabetics have a lifetime risk of 15-25% of developing a DFU1, which can lead to significant decreases in the quality of life, limitations in mobility, function and independence, and increased chance of depression and anxiety. In addition, diabetics post-LEA have high rates of mortality, with 30% dying in the first year post LEA and 70% at 5 years (more than the lifetime risk of dying from cancers). What differentiates a DFU that heals and one that progresses to LEA is often the vascularity of the limb; the diabetic lower extremity often becomes ischemic due to the vascular sequelae that are a common complication of diabetes, which hampers wound closure and immune clearance of wound-associated infections. Understanding limb oxygenation can direct treatment of a DFU, which may require limb revascularization to heal.

DETAILED DESCRIPTION:
The MultIspectral MObile tiSsue Assessment (MIMOSA) Imager acquires digital images to calculate anatomical details of chronic wounds (e.g. diameter, surface area, and perimeter). The device can be worn from a lanyard, and clips onto a smartphone, using natural ambient lighting to capture images of a wound. The MIMOSA also uses up to 6 near-infrared LEDs to illuminate tissue with different wavelengths of light to assess tissue oxygenation.

The Food and Drug Administration (FDA) has previously approved a near-infrared device called the Kent camera for the assessment of tissue oxygenation. The goal of this proposal is to assess tissue oxygenation in a group of healthy volunteers with both the MIMOSA near-infrared imaging device and the Kent Camera.

The investigators hope to show that the MIMOSA Imager is substantially equivalent to the Kent Camera, and as such, the investigators are modeling the investigator's experiments on data previously published by the makers of the Kent Camera. The MIMOSA Imager is a contact-less device, and differs from the Kent Camera only in that it is smaller and more portable.

ELIGIBILITY:
Inclusion Criteria:

Age (years) 26 ± 3 (22-33) Gender (male/female) 6/6 Height (m) 1.70 ± 0.10 (1.56-1.83) Weight (kg) 65 ± 11 (49-79) Body mass index (kg/m2) 22 ± 2 (20-26) Systolic pressure (mmHg) 115 ± 15 (83-138) Diastolic pressure (mmHg) 73 ± 10 (59-91)

Exclusion Criteria:

1. Health concerns including diabetes
2. Patients who are unable to understand the aims of the study and not give informed consent

Ages: 22 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers will be recruited at St. Michael's Hospital including staff. The following inclusion criteria will be strictly followed:
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Tissue oxygenation is detected on both the MIMOSA Imager and Kent camera. | 1 year
  The MIMOSA Imager and Kent camera can both detect similar levels of tissue oxygenation.

IPD SHARING:
Plan to Share IPD: Undecided
TBD upon REB review.

REFERENCES:
- [Background] Pelletier C, Dai S, Roberts KC, Bienek A, Onysko J, Pelletier L. Report summary. Diabetes in Canada: facts and figures from a public health perspective. Chronic Dis Inj Can. 2012 Dec;33(1):53-4. PMID 23294922
- [Background] V. Hartwig, M. Marinelli, F. Rocco, and A. L'Abbate, "Assessment of Microvascular Function Using Near-Infrared Spectroscopic 2D Imaging of Whole Hand Combined with Vascular Occlusion Test," J. Med. Biol. Eng., vol. 36, no. 1, pp. 87-95, Feb. 2016.
- [Background] Skrepnek GH, Mills JL Sr, Armstrong DG. A Diabetic Emergency One Million Feet Long: Disparities and Burdens of Illness among Diabetic Foot Ulcer Cases within Emergency Departments in the United States, 2006-2010. PLoS One. 2015 Aug 6;10(8):e0134914. doi: 10.1371/journal.pone.0134914. eCollection 2015. PMID 26248037
- [Background] Serrano V, Spencer-Bonilla G, Boehmer KR, Montori VM. Minimally Disruptive Medicine for Patients with Diabetes. Curr Diab Rep. 2017 Sep 23;17(11):104. doi: 10.1007/s11892-017-0935-7. PMID 28942581
- [Background] Cross KM, Leonardi L, Payette JR, Gomez M, Levasseur MA, Schattka BJ, Sowa MG, Fish JS. Clinical utilization of near-infrared spectroscopy devices for burn depth assessment. Wound Repair Regen. 2007 May-Jun;15(3):332-40. doi: 10.1111/j.1524-475X.2007.00235.x. PMID 17537120
- [Background] Leung G, Duta D, Perry J, Leonardi L, Fish J, Cross K. Rapid tissue viability evaluation using methemoglobin as a biomarker in burns. Int J Burns Trauma. 2018 Oct 20;8(5):126-134. eCollection 2018. PMID 30515351
- [Background] Vashist SK, Schneider EM, Luong JH. Commercial Smartphone-Based Devices and Smart Applications for Personalized Healthcare Monitoring and Management. Diagnostics (Basel). 2014 Aug 18;4(3):104-28. doi: 10.3390/diagnostics4030104. PMID 26852680
- [Background] Corser W, Xu Y. Facilitating patients' diabetes self-management: a primary care intervention framework. J Nurs Care Qual. 2009 Apr-Jun;24(2):172-8. doi: 10.1097/01.NCQ.0000347456.59289.22. PMID 19287258
- [Background] Griffith ML, Siminerio L, Payne T, Krall J. A Shared Decision-Making Approach to Telemedicine: Engaging Rural Patients in Glycemic Management. J Clin Med. 2016 Nov 17;5(11):103. doi: 10.3390/jcm5110103. PMID 27869655
- [Background] Bonoto BC, de Araujo VE, Godoi IP, de Lemos LL, Godman B, Bennie M, Diniz LM, Junior AA. Efficacy of Mobile Apps to Support the Care of Patients With Diabetes Mellitus: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. JMIR Mhealth Uhealth. 2017 Mar 1;5(3):e4. doi: 10.2196/mhealth.6309. PMID 28249834